CLINICAL TRIAL: NCT01602939
Title: Subcutaneous Cladribine Plus Pegylated Interpheron Alfa-2a in Advanced Systemic Mastocytosis With D816V and Other Exon 17 KIT Mutations.
Brief Title: Cladribine Plus Pegylated Interpheron Alfa-2a in Systemic Mastocytosis
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital Virgen de la Salud (Other)
Responsible Party: Principal Investigator, LUIS ESCRIBANO, Director of the Instituto de Estudios de Mastocitosis de Castilla La Mancha, Hospital Virgen de la Salud
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EC11-187
Record Dates: First submitted 2012-05-16; First posted 2012-05-21 (Estimated); Last update posted 2016-08-29 (Estimated); Status verified 2016-08

CONDITIONS: Systemic Mastocytosis
Keywords: Mast cell; Mastocytosis; Mast cell disease
MeSH Terms: conditions — Mastocytosis, Systemic; Mastocytosis; Mast Cell Activation Disorders | interventions — Cladribine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 2CDA+IFN (Experimental)
  Interventions: Drug: Cladribine and pegylated interpheron alpha-2a

INTERVENTIONS:
Drug: Cladribine and pegylated interpheron alpha-2a — Cladribine (0.07 mg/Kg/day) s.c for 5 consecutive days each month for a total of 6 months.Cladribine daily doses could be increased up to 0.14 mg/Kg in the fourth, fifth and sixth cycles of therapy if no objetive response is achieved after the third cycle.
  Pegylated Interpheron alpha-2a (1 mcgr/Kg) s.c weekly for a total of 6 months.

SUMMARY:
The aim of this study is to evaluate the efficacy in terms of clinical and biological response rates of Cladribine plus Pegylated Interpheron alpha-2a therapy in patients with advanced systemic mastocytosis carrying D816V or other exon 17 KIT mutations.

ELIGIBILITY:
Inclusion Criteria:

* Age older than 18 years.
* Diagnosis of advanced systemic mastocytosis (aggressive systemic mastocytosis or proggressing systemic mastocytosis) with D816V or other exon 17 KIT mutations.
* ECOG ≤ 3.
* Signed informed consent.

Exclusion Criteria:

* Impaired liver function (total bilirubin ≥ 2.0 mg/dl, AST or ALT > 3 x upper limit of normal)not related to mastocytosis.
* Impaired renal function (≥ 2.0 mg/dL)not related to mastocytosis.
* Grade III-IV cytopenias not related to mastocytosis. Severe cardiopathy (grade III/IV of NYHA, or left ventricular ejection fraction < 50%).
* Pregnancy or breastfeeding.
* Female patients who do not use contraceptive methods.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2012-05; Primary Completion 2017-02 (Estimated); Study Completion 2017-06 (Estimated)

PRIMARY OUTCOMES:
To evaluate the effect of therapy on bone marrow mast cell infiltration. | 6 months
  Evaluation of bone marrow response will be assessed by immunohistochemestry, citology, flow cytometry and molecular analyses of bone marrow samples.

SECONDARY OUTCOMES:
To determine the effect of therapy on serum tryptase levels and other altered peripheral blood parameters due to mastocytosis. | 6 months
  Serum tryptase and any other mastocytosis-related altered biochemical parameter at diagnosis will be measured monthly until the end of therapy.
To evaluate the effect of therapy on mast cell-mediator release symptoms: pruritus, flushing, gastrointestinal symptoms or anaphylaxis). | 6 months
  Specific questionnaires regarding mast cell-mediator release symptoms will be filled monthly by each patient until the end of therapy.
To determine de safety of combined therapy with low doses of cladribine plus pegylated interpheron alpha-2a. | 6 months
  Potentially drugs-related adverse events will be recorded in each case following accepted criteria (NIH CTCAE).
To evaluate the effect of therapy on mastocytosis skin lesions. | 6 moths
  Evaluation of cutaneous response will be assessed by macroscopic inspection including photographs and by skin immunohistochemestry.
To evaluate the effect of therapy on mastocytosis-related organomegalies. | 6 months
  Evaluation of organomegalies response will be assessed by abdominal ultrasound and/or computerized tomography.
To evaluate the effect of therapy on mastocytosis-related bone alterations. | 6 months
  Evaluation of bone response will be assessed by X-ray survey and/or computerized tomography.

CONTACTS AND LOCATIONS:
Overall Officials: Luis Escribano, MD, PhD, Principal Investigator — Instituto de Estudios de Mastocitosis de Castilla La Mancha
Locations (1):
- Instituto de Estudios de Mastocitosis de Castilla La Mancha; Hospital Virgen del Valle, Toledo, Toledo, Spain

IPD SHARING:
Plan to Share IPD: Undecided